CLINICAL TRIAL: NCT06371859
Title: Human-AI Collaborative Intelligence for Improving Fetal Flow Management: A Randomized Trial
Brief Title: Human-AI Collaborative Intelligence for Improving Fetal Flow Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Slagelse Hospital (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Zahra Bashir, Ph.d.student, medical doctor and primary investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 3-3031-2915/1
Record Dates: First submitted 2023-05-09; First posted 2024-04-17 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes will be used and opened at the time of inclusion of each participant. Each participant will be randomized to either AI support or no support. The allocation of participants will be performed by (XYZ) who does not have access to the randomization order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "XAI feedback on MCA/UA Doppler spectral curves and gate placement suggestions" (Experimental): The XAI feedback group will place a gate on MCA/UA images and evaluate the Doppler spectrum with AI feedback.
  N=46 clinicians (Clinicians will be divided into two groups (XAI feedback & No XAI feedback groups) of 46 each, matched for experience levels across hospitals)
  Interventions: Behavioral: "XAI feedback on MCA/UA Doppler spectral curves and gate placement suggestions"
- "No XAI feedback" (No Intervention): The control group will place a gate on MCA/UA images and evaluate the Doppler spectrum without AI feedback.
  N=46 clinicians (Clinicians will be divided into two groups (XAI feedback & No XAI feedback groups) of 46 each, matched for experience levels across hospitals)

INTERVENTIONS:
Behavioral: "XAI feedback on MCA/UA Doppler spectral curves and gate placement suggestions" — This study includes 1840 ultrasound images, split into UA and MCA flow and spectrum images, each duplicated for a total of 3680 images to compare explainable AI (XAI) feedback vs. no feedback. The investigators will provide matched sets of 40 images (one for the XAI group and one for the non-XAI group) to participants. Participants are matched based on their level of experience within each hospital (Resident physicians, obstetricians, and gynecologists with obstetric ultrasound experience).
  All participants are instructed to place gates on the flow images of the umbilical artery and the middle cerebral artery and to assess the quality of the resulting flow curves. Specifically, for flow images, participants must identify the most appropriate gate placement. For spectral flow curves, they are to decide if the curves are of sufficient quality to guide medical management decisions.
  Arms: "XAI feedback on MCA/UA Doppler spectral curves and gate placement suggestions"

SUMMARY:
This randomized controlled study evaluates the effectiveness of explainable AI (XAI) in improving clinicians' interpretation of Doppler ultrasound images (UA and MCA) in obstetrics. It involves 92 clinicians, randomized into intervention and control groups. The intervention group receives XAI feedback, aiming to enhance accuracy in ultrasound interpretation and medical decision-making.

Objectives:

1. To develop an interpretable model for commonly used Doppler flows, specifically the Pulsatility Index (PI) of the umbilical artery (UA) and middle cerebral artery (MCA), with the aim to provide quality feedback on Doppler spectrum images and suggest potential gate placements.
2. To test the effects of providing Explainable AI (XAI)-feedback for clinicians compared with no feedback on their accuracy in ultrasound interpretation and management.

DETAILED DESCRIPTION:
Currently, Doppler ultrasound velocimetry serves as a crucial tool in obstetric practice, particularly for assessing the umbilical artery (UA) and middle cerebral artery (MCA) in uteroplacental-fetal circulation. While Doppler ultrasound is valuable for detecting conditions like fetal anemia and placental insufficiency, its accuracy relies on operator expertise. Artificial intelligence (AI) offers potential enhancements, especially in high-risk pregnancies. However, existing AI applications in fetal ultrasound often lack transparency, leading to user distrust. This study aims to address these limitations by developing an explainable AI model to assist clinicians in interpreting Doppler ultrasound images of UA and MCA for improved management of high-risk pregnancies.

The study's objectives are:

1. To develop an interpretable model for commonly used Doppler flows, specifically the Pulsatility Index (PI) of the umbilical artery (UA) and middle cerebral artery (MCA), with the aim to provide quality feedback on Doppler spectrum images and suggest potential gate placements.
2. To test the effects of providing Explainable AI (XAI)-feedback for clinicians compared with no feedback on their accuracy in ultrasound interpretation and management.

All participants will be instructed to provide gate placement for flow images of the umbilical artery and the MCA, and to evaluate the quality of the resulting flow curves. Each participant will be required to evaluate a total of 40 unique images (10 flow images for UA and MCA, 10 spectral doppler images for UA and MCA, respectively). From the four groups (UA-flow, UA-spectrum, MCA-flow & MCA-spectrum) the investigators will provide matched sets of 40 images that are provided to participants, who are matched for their level of experience within each hospital (PGY 1-2; PGY 3-5; board certified Obstetricians). For flow images, the participants will be instructed to identify the most appropriate gate placement. For the spectral flow curves, participants will be asked to evaluate whether the flow curves were of sufficient quality to inform medical management decisions.

The inclusions criteria for MCA and UA images will be images taken from the third trimester (>= week 28).

Study Design: Randomized controlled trial

Data Source: 1840 unique ultrasound scans including umbilical artery (UA) and middle cerebral artery (MCA) measurements. The 1840 unique images includes: 460 images of UA-flow images, 460 UA-spectrum images, 460 MCA-flow images and 460 MCA-spectrum images.

Participants: 92 clinicians with varying competence levels across four different university hospitals.

Intervention: XAI feedback on MCA/UA Doppler spectral curves and gate placement suggestions.

Control Group: No XAI feedback.

Procedure: Clinicians will be divided into two groups of 46 each, matched for experience levels across hospitals. The control group will place a gate on MCA/UA images and evaluate the Doppler spectrum without AI feedback, while the intervention group will perform the same tasks with access to AI feedback.

Outcome Measures: The participants' responses in the two groups are reviewed by two fetal medicine sonographers who evaluate the participants' answers independently of each other. In a disagreement, the two sonographers reach a consensus after discussion.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion is the use of ultrasound at least once per week

Exclusion Criteria:

* The exclusion criterion is the absence of experience in ultrasound scanning.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Responses will be reviewed independently by two fetal medicine sonographers, and in case of disagreement between the two experts, a consensus will be reached. | 1 months
  The accuracy in each group (AI-feedback and without AI-feedback group) was defined as the percentage difference in the number of correctly managed flow images between the two groups, assessed by two fetal medicine sonographers.
  Correct management was defined as: Correct gate placement (multiple sites possible) AND Correct identification of flow curves that were of adequate quality to allow medical decision-making.

SECONDARY OUTCOMES:
Accuracy of flow image management among competence groups | 1 months
  The secondary outcome is to categorize participants into competence groups (trainees, obstetricians, and gynecologists with obstetric experience) and then examine the percentage difference in the accuracy of flow image management among these competence groups within both the AI-feedback and the non-AI-feedback groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region of Denmark
  - Slagelse Hospital, Slagelse, Region Sjælland